CLINICAL TRIAL: NCT03768401
Title: Accessible Mobile Health and Wellness
Acronym: CHAMPs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding/grant expired.
Sponsor: Kristin Zhao, PhD (Other)
Collaborators: Southeastern Minnesota Center for Independent Living (Unknown)
Responsible Party: Sponsor-Investigator, Kristin Zhao, PhD, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-008524
Record Dates: First submitted 2018-07-17; First posted 2018-12-07 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Physical Disability; Neurologic Dysfunction
MeSH Terms: conditions — Neurologic Manifestations | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Seminars and Wellness Clinics (Experimental): I. Community outreach educational seminars about wellness and exercise while living with a neurological physical disability and measurement of the effects of these seminars for training individuals with neurological physical disabilities and their care givers (family, therapists, community personal trainers and community funders such as Lions or Rotary Clubs) about how to create a safe cost-effective exercise program .
  II. Creation and measurement of the effects of a wellness clinic for those with a neurological physical disability.
  Interventions: Other: Education; Behavioral: Trial Exercise Modalities

INTERVENTIONS:
Other: Education — Seminars about wellness and exercise, and resulting therapeutic programs, while living with a neurological physical disability.
Behavioral: Trial Exercise Modalities — Wellness/exercise clinics located at Mayo Clinic, Rochester will be offered to persons with neurological physical disabilities on a regular basis, at least monthly, during the last half of the trial period.

SUMMARY:
Can community outreach education help develop self-sustaining wellness and exercise programs, and will associated wellness clinics help persons with a neurological physical disability achieve better well-being?

ELIGIBILITY:
Inclusion Criteria:

* [for community participants/caregivers/family members] Ability to demonstrate clear communication and understanding of English.
* [for participants with neurological physical conditions] Neurological physical conditions including cerebral palsy, spinal cord injury, stroke, multiple sclerosis, or similar diagnoses
* [for educational seminars] > 6 years of age.
* [for wellness/exercise clinic] 18 65 years of age
* [for wellness/exercise clinic; participants with neurological physical conditions] Clearance by primary care or treating physician

Exclusion Criteria:

* [for participants with neurological physical conditions] Unstable fractures
* [for participants with neurological physical conditions] Uncontrolled hypertension (combined systolic/diastolic > 140/90 mmHg)
* [for participants with neurological physical conditions] Enrollment of individual deemed by study staff to be unsafe

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Incidence of new self-sustaining wellness and exercise programs | 3 months post end of wellness clinics
  Incidence of new self-sustaining wellness and exercise programs, as determined by Follow-up Site Staff Survey

SECONDARY OUTCOMES:
Efficacy of seminars for individuals with a neurological physical disability | 3 months post end of wellness clinics
  Efficacy of seminars, as determined by repeated t-tests based on the Exercise Self-Efficacy Survey (ESES), a 10-question survey with scores of 1 to 4 (with 4 being the best outcome), summed for a minimum score of 10, and a maximum score of 40.
Efficacy of seminars for caregivers and clinic staff of patients with neurological physical disabilities | 3 months post end of wellness clinics
  Efficacy of seminars, as determined by repeated t-tests based on the Exercise Efficacy for Caregivers and Staff, a 10-question survey with scores of 1 to 4 (with 4 being the best outcome), summed for a minimum score of 10, and a maximum score of 40.
Efficacy of wellness clinics | 3 months post end of wellness clinics
  Efficacy of wellness clinics, as determined by repeated t-tests

CONTACTS AND LOCATIONS:
Overall Officials: Kristin D Zhao, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials